CLINICAL TRIAL: NCT05927792
Title: Efficacy and Mechanism of Repetitive Transcranial Magnetic Stimulation in Children With Autism Spectrum Disorders: a Multicenter, Randomized Controlled Trial
Brief Title: Efficacy and Mechanism of Repetitive Transcranial Magnetic Stimulation in Children With Autism Spectrum Disorders
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Mental Health Center (Other); Zhengzhou Children's Hospital, China (Other); Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Fei Li, Chief Physician ,Doctoral Supervisor, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XHEC-C-2023-043
Record Dates: First submitted 2023-06-13; First posted 2023-07-03 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Autism Spectrum Disorder
Keywords: Repetitive Transcranial Magnetic Stimulation（rTMS）; Autism Spectrum Disorder; Intervention; Social Deficits; Language Function; Children
MeSH Terms: conditions — Autism Spectrum Disorder; Language

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants, their legal guardians, and the assessors were unaware of the grouping except for the intervention operator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): participants in intervention group will receive accelerated continuous theta-burst stimulation (a-cTBS) on the left primary motor cortex (M1) for 5 consecutive days.
  Interventions: Device: repeated transcranial magnetic stimulation (continuous theta-burst stimulation)
- Sham Group (Sham Comparator): The sham group will be stimulated with a pseudo-stimulation coil, which emitted sounds with the same intensity, rhythm and vibratory sensation as the real stimulation, and the intervention target, duration and frequency are the same as the real intervention group.
  Interventions: Device: sham repeated transcranial magnetic stimulation

INTERVENTIONS:
Device: repeated transcranial magnetic stimulation (continuous theta-burst stimulation) — Participants in intervention group will receive cTBS over the left M1for 5 consecutive days. The detailed parameters as follows: 80% of resting motor threshold (RMT), 60 cycles of 10 bursts of three pulses at 50 Hz were delivered in 2-second trains (5 Hz) with no intertrain interval (i.e. triplet standard cTBS, 1800 pulses, 120s). Stimulation sessions were delivered hourly, 10 sessions were applied per day (18,000 pulses/day).
  Arms: Intervention Group
Device: sham repeated transcranial magnetic stimulation — The sham group will be stimulated with a pseudo-stimulation coil, which emitted sounds with the same intensity, rhythm and vibratory sensation as the real stimulation, and the intervention target, duration and frequency are the same as the real intervention group.
  Arms: Sham Group

SUMMARY:
This study is a prospective, multicenter, randomized, single-blind controlled trial to enroll 200 children with autism spectrum disorders (ASD). The investigators hope to further explore the effectiveness of accelerated continuous theta-burst stimulation (a-cTBS) over the left primary motor cortex (M1) to improve core symptoms in ASD children based on a previous open-label clinical trial.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, randomized, single-blind controlled trial. Shanghai Xinhua hospital, Qilu hospital and Zhengzhou Children's hospital expect to enroll a total of 200 children with autism spectrum disorders (ASD) to participate in this trial.

The children seen at Department of Developmental Behavioral Child Health, who meet the The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition(DSM-5) ASD diagnostic criteria and strict inclusion/exclusion criteria, can be enrolled for the intervention after informed consent.

At each study center, participants will be randomized into intervention group and sham group stratified by IQ level. The participants, their legal guardians, and the assessors were unaware of the grouping except for the intervention operator (single-blind).

During the trial, participants in intervention group will receive accelerated continuous theta-burst stimulation (a-cTBS) on the left primary motor cortex (M1) for 5 consecutive days. The sham group will be stimulated with a pseudo-stimulation coil, which emitted sounds with the same intensity, rhythm and vibratory sensation as the real stimulation, and the intervention target, duration and frequency are the same as the real intervention group.

All participants need to complete clinical assessments within 2 weeks before the cTBS intervention (pre-cTBS), repeated within 3 days after the completion of the cTBS course (post-cTBS) and 1 month following the last cTBS session (one month follow-up), respectively.

The investigators hope to further explore the effectiveness of accelerated continuous theta-burst stimulation (a-cTBS) over the left primary motor cortex (M1) to improve core symptoms in ASD children based on a previous open-label clinical trial and investigate the appropriate intervention model, effective adaptation population and underlying neurological mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4-10 years old
* Meet the diagnostic criteria for ASD of the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)
* ASD Diagnosis confirmed by the Autism Diagnostic Observation Schedule (ADOS) or Autism Diagnostic Interview, Revised (ADI-R)
* IQ of 50 or above
* Provide written informed consents

Exclusion Criteria:

* With metal implants in the body
* History of epilepsy or other neurological disease
* Require surgical treatment due to structural abnormalities indicated by brain MRI
* Diagnosed with genetic and chromosomal abnormalities
* With psychiatric/mental disorder (e.g., very early-onset schizophrenia) other than ASD
* Suffer from serious heart disease and/or severe hearing impairment
* Intracranial hypertension
* Participating in other clinical trials
* Participants who received other interventions within 4 weeks prior to enrollment.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Changes of Social Responsiveness Scale, Second Edition (SRS-2) scores from pre-intervention to post-intervention | within 2 weeks before the intervention (pre-intervention), within 3 days after the completion of the intervention course (post-intervention)
  SRS provides the multi-dimensional measure of social interaction allowing the rating of social impairment in ASD. SRS generates a total score and five theoretical subscale scores (labeled social awareness, social cognition, social communication, social motivation, restricted interests and repetitive behavior), and higher scores are indicative of greater social impairment.
Changes of Social Responsiveness Scale, Second Edition (SRS-2) scores from pre-intervention to 1 month follow-up | within 2 weeks before the intervention (pre-intervention), 1 month following the last intervention session (one month follow-up)
  SRS provides the multi-dimensional measure of social interaction allowing the rating of social impairment in ASD. SRS generates a total score and five theoretical subscale scores (labeled social awareness, social cognition, social communication, social motivation, restricted interests and repetitive behavior), and higher scores are indicative of greater social impairment.

SECONDARY OUTCOMES:
Chinese Communicative Development Inventory (CCDI) | within 2 weeks before the intervention (pre-intervention), 1 month following the last intervention session (one month follow-up)
  a parent questionnaire serves as a powerful tool to evaluate the early vocabulary development and language skills of older children with developmental disorders and the effectiveness of their interventions. CCDI yields two subscale scores, including words produced score and sentence complexity score.Higher scores suggest better language level.
Language Comprehension Test | within 2 weeks before the intervention (pre-intervention), 1 month following the last intervention session (one month follow-up)
  Peabody Picture Vocabulary Test (PPVT) is a standard assessment tool for measuring single-word comprehension, to objectively evaluate the language ability of the children involved in our study. Higher scores suggest better language level.
  Meanwhile, a sentence-picture matching test will be administered to test children's language comprehension abilities in the syntactic domain.
Multilingual Assessment Instrument for Narratives (MAIN) | within 2 weeks before the intervention (pre-intervention), 1 month following the last intervention session (one month follow-up)
  assess narrative comprehension and production skills of children who exhibited a certain level of expressive ability (at least can use flexible phrases).In this test, children tell or retell the stories and answer some questions, with assessors evaluating performance across four dimensions: story structure, structural complexity, internal state terms, and comprehension questions. Higher scores suggest better language level.
Clinical Global Impression Scale (CGI) | within 3 days after the completion of the intervention course (post-intervention), 1 month following the last intervention session (one month follow-up)
  we used CGI-I to rate how much the patient's illness has improved or worsened relative to a baseline measurement (a seven-point scale: 1 = "very much improved" to 7 = "very much worse")
Vineland Adaptive Behavior Scales, Third Edition (Vineland-3) | within 2 weeks before the intervention (pre-intervention), 1 month following the last intervention session (one month follow-up)
  The Vineland Adaptive Behavior Scales were designed to address adaptive behavior, or the personal and social skills necessary for everyday independent living. For individuals with ASDs, the Vineland can be used for tracking and reporting progress of intervention or treatment. Domains of adaptive functioning assessed with the Vineland include: Communication, Daily Living Skills, Socialization, Motor Skills. The higher scores suggest better adaptive level.
Electroencephalography (EEG) | within 2 weeks before the intervention (pre-intervention), within 2 days after the completion of the intervention course (post-intervention)
  Electroencephalography (EEG): We plan to collect resting-state and task-related EEG data from children with ASD at baseline, after 5 days of intervention after intervention to evaluate changes in power spectrum and inter-trial phase coherence (ITPC) in the alpha and theta frequency bands at different time points. The EEG data will be collected using a 128-channel EEG system with a sampling rate of 1000 Hz and a reference electrode at Cz (central zero). Prior to data collection, we will ensure that the resistance of each channel is below 100 kΩ.

CONTACTS AND LOCATIONS:
Overall Officials: Fei Li, MD, PhD, Principal Investigator — Shanghai Jiaotong University School of Medicine Xinhua Hospital
Locations (3):
- China (3):
  - Henan Children's Hospital, Zhengzhou, Henan
  - Qilu Hospital of Shandong University, Qilu, Shandong
  - Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No
Study Protocol, Statistical Analysis Plan, Informed Consent Form (ICF), etc are available through contacting researchers if required.